CLINICAL TRIAL: NCT02562560
Title: Neuropsycholgy and Neuroimaging in Transient Global Amnesia
Acronym: 2NIA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no more patient
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: 2007-A00910-53
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2015-11

CONDITIONS: Transient Global Amnesia (TGA)
MeSH Terms: conditions — Amnesia, Transient Global | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TGA (Experimental)
  Interventions: Behavioral: Neuropsychological tests; Device: Cerebral imaging (MRI, PET-FDG)
- Controls (Experimental)
  Interventions: Behavioral: Neuropsychological tests; Device: Cerebral imaging (MRI, PET-FDG)

INTERVENTIONS:
Behavioral: Neuropsychological tests
Device: Cerebral imaging (MRI, PET-FDG)

SUMMARY:
The purpose of this study is to establish a diagnosis in transient global amnesia (TGA) in assessing three episodic memory's abilities (mental simulation throught the future, and the past, the learning of personnal actions i-e the enactment effect). Secondary goal is to describe the neuronal substrates associated to the alteration of theses abilites in TGA.

ELIGIBILITY:
Inclusion Criteria:

* All the participants

  * Minimum of 7 years of education
  * French native speaker
* Healthy subjects : Non pathological Dementia rating scale score
* Patients : Clinical diagnosis of TGA according to Hodges and Warlow's criterion

Exclusion Criteria:

* Chronic neurological disease
* Encephalitis
* Endocrinal disease
* Hepatic disease
* Case history of head injury with loss of consciousness of more than one hour
* Case history of stroke
* Case history of cancer during the five last years except squamous cell carcinomas
* Alcoholism or drug addiction
* Major psychiatric disorders according the Diagnostic and Statistical Manual of -Mental Disorders

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Episodic memory scores | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Viader, PUPH, Principal Investigator — University Hospital, Caen